CLINICAL TRIAL: NCT00726167
Title: Clinical Utility of Serum Procalcitonin in the Management of Ventilator-Associated Pneumonia
Brief Title: Serum Procalcitonin Study in the Management of Ventilated Patients
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 1106537
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator associated Pneumonia; mechanically ventilated; procalcitonin; pneumonia scores
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Procalcitonin Level — Procalcitonin concentrations will be determined every day and will be compared with the clinical diagnosis based upon standard clinical practice. All subjects enrolled will be followed until the patient is either extubated or discharged from the SICU.
  Other Names: PCT

SUMMARY:
The purpose of this study is to test a new method for diagnosing and monitoring Ventilator-Associated Pneumonia, which is a major killer among ICU patients. The method requires analysis of a small amount of the patient's blood for concentration of a hormone called Procalcitonin.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia is a leading cause of mortality in critically ill patients. The purpose of this study is to evaluate the relationship between the onset/progress/resolution of pneumonia and the levels of Procalcitonin, a prohormone whose concentrations fluctuate in response to bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Are willing to give or who's proxy is willing to consent to be a study subject
* Are at least 18 years of age;
* Who are mechanically ventilated surgical intensive care unit patients.

Exclusion Criteria:

* Participation in any investigational device or drug trial within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated surgical intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Correlation of Procalcitonin concentration with the LungGuardian-derived Pneumonia Score in mechanically ventilated surgical intensive care unit patients. Using the data collected a positive and negative predictive value will be calculated. | Once daily

SECONDARY OUTCOMES:
antibiotic status (appropriateness, effectiveness, discontinuation criteria) | Once daily
intubation date | Once daily
microbiology data | Once daily
PCT levels | Once daily
pneumonia-related symptoms (including tracheal secretion character, body temperature, oxygenation, and WBC counts) | Once daily

CONTACTS AND LOCATIONS:
Overall Officials: Jerry B Rogers, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fartoukh M, Maitre B, Honore S, Cerf C, Zahar JR, Brun-Buisson C. Diagnosing pneumonia during mechanical ventilation: the clinical pulmonary infection score revisited. Am J Respir Crit Care Med. 2003 Jul 15;168(2):173-9. doi: 10.1164/rccm.200212-1449OC. Epub 2003 May 8. PMID 12738607
- [Background] Christ-Crain M, Muller B. Procalcitonin and pneumonia: is it a useful marker? Curr Infect Dis Rep. 2007 May;9(3):233-40. doi: 10.1007/s11908-007-0037-9. PMID 17430706
- [Background] Christ-Crain M, Muller B. Procalcitonin in bacterial infections--hype, hope, more or less? Swiss Med Wkly. 2005 Aug 6;135(31-32):451-60. doi: 10.4414/smw.2005.11169. PMID 16208582
- [Background] Ibrahim EH, Tracy L, Hill C, Fraser VJ, Kollef MH. The occurrence of ventilator-associated pneumonia in a community hospital: risk factors and clinical outcomes. Chest. 2001 Aug;120(2):555-61. doi: 10.1378/chest.120.2.555. PMID 11502658
- [Background] Rello J, Ollendorf DA, Oster G, Vera-Llonch M, Bellm L, Redman R, Kollef MH; VAP Outcomes Scientific Advisory Group. Epidemiology and outcomes of ventilator-associated pneumonia in a large US database. Chest. 2002 Dec;122(6):2115-21. doi: 10.1378/chest.122.6.2115. PMID 12475855
- [Background] Tablan OC, Anderson LJ, Besser R, Bridges C, Hajjeh R; CDC; Healthcare Infection Control Practices Advisory Committee. Guidelines for preventing health-care--associated pneumonia, 2003: recommendations of CDC and the Healthcare Infection Control Practices Advisory Committee. MMWR Recomm Rep. 2004 Mar 26;53(RR-3):1-36. PMID 15048056
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Nylen E, Muller B, Becker KL, Snider R. The future diagnostic role of procalcitonin levels: the need for improved sensitivity. Clin Infect Dis. 2003 Mar 15;36(6):823-4; author reply 826-7. doi: 10.1086/368088. No abstract available. PMID 12627371
- [Background] Mueller B and Prat C. Markers in acute inflammation in assessing and managing lower respiratory tract infections; focus on procalcitonin. Clin Microbiol Infect 2006; 12(Suppl):8-16
- [Background] Phillips JO, Metzler MH, Huckfeldt RE, Keller ME, McBride CL. A Prospective evaluation of a simple disease management plan for nosocomial pneumonia in the ventilated trauma patient. Crit Care Med 1999: 27: 143